CLINICAL TRIAL: NCT05299216
Title: Effect of Conventional Physical Therapy With or Without Diaphragm Manual Therapy in Patients With Chronic Non-Specific Low Back Pain
Brief Title: Effect of Diaphragm Manual Therapy With Conventional Physical Therapy in Chronic Non-Specific Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, M. Ammar Ahmad Sohail, Principal Investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRMAAS
Record Dates: First submitted 2022-03-04; First posted 2022-03-28 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain; Chronic Low-back Pain
Keywords: Low Back Pain, Manual Therapy, Conventional Physical Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive Manual Diaphragm Technique in addition to Conventional Physical Therapy. Treatment will be provided for a total of four weeks, thrice a week.
  Interventions: Other: Manual Diaphragm Technique; Other: Conventional Physical Therapy
- Group B (Active Comparator): Group B will receive Conventional Physical Therapy and Sham Diaphragm Technique. Conventional Physical Therapy group comprises electrotherapeutic treatment and exercise plan. Treatment will be provided for a total of four weeks, thrice a week.
  Interventions: Other: Conventional Physical Therapy; Other: Sham Diaphragm Manual Technique

INTERVENTIONS:
Other: Manual Diaphragm Technique — Treatment group will receive Manual Diaphragm Technique in addition to Conventional Physical Therapy. Therapist will make physical contact to the underside of the 7th to 10th rib costal cartilages. During the inspiratory phase, the therapist will use both hands to gently pull the points of contact in the direction of the head. During exhalation, the therapist will maintain resistance. The procedure will be done in two sets of ten deep breaths, separated by a one-minute pause.
  Arms: Group A
Other: Conventional Physical Therapy — Conventional Physical Therapy group comprises electrotherapeutic treatment and exercise plan. Subjects will undergo a thermal continuous ultrasound, conventional transcutaneous electrical nerve stimulation and a hot pack.
  Stretching activities for the back, iliopsoas, and hamstring muscles, as well as abdominal muscle strengthening exercises, will be included in the workout.
Other: Sham Diaphragm Manual Technique — The Control group will also receive a sham diaphragm release technique. The therapist and participant will have the same manual contacts, duration, and placement as the treatment group, but the therapist will simply use a light touch with the same anatomical landmarks and will not apply pressure.
  Arms: Group B

SUMMARY:
A randomized single-blind clinical study will be performed. A sample size of 34 patients including only male gender, will be taken from various clinical settings of Faisalabad. Non-probability purposive sampling technique will be used. Patients will be randomly allocated into two groups. Treatment Group A will perform Conventional Physical Therapy and Diaphragm Manual Therapy and Group B will perform Conventional Physical Therapy and Sham Diaphragm Manual Therapy. Numerical Pain Rating Scale and lumbar range of motion scores will be assessed at pre-treatment, 2nd-week post-treatment and 4th-week post-treatment. Oswestry Disability Index scores and Short Form 12 Health Survey Questionnaire will be assessed at pre-treatment and 4th-week post-treatment. Statistical analysis will be performed on Statistical Package for the Social Sciences Version 25.

DETAILED DESCRIPTION:
Over 80% of people experience Lower back pain in their lives, of which 23% suffer from chronic pain. Physiotherapists use multiple treatment options for treating non-specific chronic low back pain such as joint mobilization, therapeutic exercises, electrotherapeutic modalities and soft tissue release techniques.

The objective of the study is to determine the effect of conventional physical therapy with or without diaphragm manual therapy in patients with chronic non-specific low back pain.

A randomized, single-blind clinical study will be performed. A sample size of 34 patients comprising of only male gender will be taken from various clinical settings of Faisalabad. Non-probability purposive sampling technique will be used. Patients will be randomly allocated into two groups. Treatment Group A will perform Conventional Physical Therapy and Diaphragm Manual Therapy and Group B will perform Conventional Physical Therapy and Sham Diaphragm Manual Therapy. Numerical Pain Rating Scale and lumbar range of motion scores will be assessed at pre-treatment, 2nd-week post-treatment and 4th-week post-treatment. Oswestry Disability Index scores and Short Form 12 Health Survey Questionnaire will be assessed at pre-treatment and 4th-week post-treatment.

Statistical analysis will be performed on Statistical Package for the Social Sciences Version 25. Mean ± Standard Deviation will be used to present Quantitative variables while Qualitative variables will be shown through frequency tables and percentages will be shown in the form of frequency tables and percentages. Summary of group measurements will be represented through Graphs. Normal distribution of data will be analyzed through skewness, kurtosis and Shapiro wilk test. If data is found normally distributed, then parametric tests will be applied, which will include an Independent sample t-test for measuring inter-group changes. Paired Sample t-test/Repeated measure ANOVA for measuring intra-group differences. If data is found non-normally distributed, then non-parametric tests will be applied, which will include Mann-Whitney U-Test for measuring inter-group changes and Wilcoxon Test/Friedman Test for measuring intra-group differences. P-value ≤ 0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-55 years.
* Male gender
* Patients diagnosed as having non-specific chronic low back pain from the last 12 weeks minimum.
* Pain rating of at least 3 on Numerical Pain Rating Scale.

Exclusion Criteria:

* Previous history of spinal trauma, fracture or surgery.
* Patients with lumbar disc herniation and radicular low back pain.
* Patients having any spinal malignancy, psychological distress, infectious disorder or systemic disorder.
* Patients with tuberculosis of the spine.
* Patients with musculoskeletal injuries of the lower extremities.
* Patients who regularly consume anti-inflammatory or analgesic drugs.
* Previous history of manual treatment in the last month.
* Patients having contraindications for manual therapy.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male Gender
Enrollment: 34 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Numerical Pain Rating Scale (Pain) | Change from baseline at 2nd week and Change from 2nd week at 4th week.
  Numerical Pain Rating Scale will be used to measure back pain. Score of scale ranges from 0 (no pain) to 10 (worst possible pain).
Change in Universal Goniometer (Lumbar Range of Motion) | Change from baseline at 2nd week and Change from 2nd week at 4th week.
  Universal Goniometer will be used to measure Lumbar Range of Motion.

SECONDARY OUTCOMES:
Change in Oswestry Disability Index (Back Function Disability) | Change from baseline at 2nd week and Change from 2nd week at 4th week.
  Oswestry Disability Index original English version (United States) and Urdu translated version (Pakistan) to measure back function disability. Score of this scale ranges from 0(no disability) to 50(completely disabled).
Change in Short Form 12 Health Survey (Health Related Quality of Life) | Change from baseline at 2nd week and Change from 2nd week at 4th week.
  Short Form 12 Health Survey Questionnaire original English version (United States) and Urdu translated version (Pakistan) will be used to assess health related quality of life. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mariam Mehmood, MS-OMPT, Principal Investigator — University of Faisalabad
Locations (2):
- Pakistan (2):
  - Muhammad Hospital, Samnabad, Faisalabad, Punjab Province
  - Physio & Pain Care Clinic, Faisalabad, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rocha T, Souza H, Brandao DC, Rattes C, Ribeiro L, Campos SL, Aliverti A, de Andrade AD. The Manual Diaphragm Release Technique improves diaphragmatic mobility, inspiratory capacity and exercise capacity in people with chronic obstructive pulmonary disease: a randomised trial. J Physiother. 2015 Oct;61(4):182-9. doi: 10.1016/j.jphys.2015.08.009. Epub 2015 Sep 19. PMID 26386894
- [Background] Ozkaraoglu DK, Tarakci D, Algun ZC. Comparison of two different electrotherapy methods in low back pain treatment. J Back Musculoskelet Rehabil. 2020;33(2):193-199. doi: 10.3233/BMR-181199. PMID 31594200
- [Background] Kachanathu SJ, Alenazi AM, Seif HE, Hafez AR, Alroumim MA. Comparison between Kinesio Taping and a Traditional Physical Therapy Program in Treatment of Nonspecific Low Back Pain. J Phys Ther Sci. 2014 Aug;26(8):1185-8. doi: 10.1589/jpts.26.1185. Epub 2014 Aug 30. PMID 25202177
- [Background] Alsufiany MB, Lohman EB, Daher NS, Gang GR, Shallan AI, Jaber HM. Non-specific chronic low back pain and physical activity: A comparison of postural control and hip muscle isometric strength: A cross-sectional study. Medicine (Baltimore). 2020 Jan;99(5):e18544. doi: 10.1097/MD.0000000000018544. PMID 32000363
- [Background] Joshi VD, Raiturker PP, Kulkarni AA. Validity and reliability of English and Marathi Oswestry Disability Index (version 2.1a) in Indian population. Spine (Phila Pa 1976). 2013 May 15;38(11):E662-8. doi: 10.1097/BRS.0b013e31828a34c3. PMID 23380824
- [Background] Amjad F, Mohseni-Bandpei MA, Gilani SA, Ahmad A, Waqas M, Hanif A. Urdu version of Oswestry disability index; a reliability and validity study. BMC Musculoskelet Disord. 2021 Mar 29;22(1):311. doi: 10.1186/s12891-021-04173-0. PMID 33781267
- [Background] Ibrahim AA, Akindele MO, Ganiyu SO, Kaka B, Abdullahi BB, Sulaiman SK, Fatoye F. The Hausa 12-item short-form health survey (SF-12): Translation, cross-cultural adaptation and validation in mixed urban and rural Nigerian populations with chronic low back pain. PLoS One. 2020 May 7;15(5):e0232223. doi: 10.1371/journal.pone.0232223. eCollection 2020. PMID 32379769
- [Background] Marti-Salvador M, Hidalgo-Moreno L, Domenech-Fernandez J, Lison JF, Arguisuelas MD. Osteopathic Manipulative Treatment Including Specific Diaphragm Techniques Improves Pain and Disability in Chronic Nonspecific Low Back Pain: A Randomized Trial. Arch Phys Med Rehabil. 2018 Sep;99(9):1720-1729. doi: 10.1016/j.apmr.2018.04.022. Epub 2018 May 19. PMID 29787734
- [Background] Comachio J, Magalhaes MO, Campos Carvalho E Silva APM, Marques AP. A cross-sectional study of associations between kinesiophobia, pain, disability, and quality of life in patients with chronic low back pain. Adv Rheumatol. 2018 Jun 22;58(1):8. doi: 10.1186/s42358-018-0011-2. PMID 30657061